CLINICAL TRIAL: NCT02708914
Title: A Phase III Trial to Compare the Safety and Efficacy of Intravenous UB-851 and Eprex® With an Extension Safety Evaluation in Subjects With Renal Anemia on Hemodialysis
Brief Title: Study to Compare the Safety and Efficacy of UB-851 and Eprex®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UBI Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P304-EPO
Record Dates: First submitted 2016-02-23; First posted 2016-03-15 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2022-05

CONDITIONS: Renal Anemia
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UB-851 (Other)
  Interventions: Biological: UB-851
- Eprex then UB-851 (Other)
  Interventions: Biological: UB-851; Biological: Eprex

INTERVENTIONS:
Biological: UB-851 — UB-851 (rhEPO) has been developed as a biosimilar product to Eprex®.
Biological: Eprex — Eprex® is chosen as the comparator.
  Arms: Eprex then UB-851

SUMMARY:
The primary objective of this study is to evaluate a 1:1 dose conversion from Eprex® to UB-851 in terms of clinical efficacy and safety in subjects with chronic renal failure receiving hemodialysis.

DETAILED DESCRIPTION:
This is a 52-week, phase III trial consisting of two parts:

Part I is designed as a double-blind, randomized, multicenter, parallel-group study to evaluate the efficacy and safety of UB-851 in comparison to Eprex® in subjects with renal anemia on hemodialysis with a treatment period of 24 weeks.

Part II is designed as a single-arm, safety evaluation period (from week 25 to week 52) to evaluate the long-term safety and immunogenicity of UB-851.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subjects signed informed consent before undergoing any study procedures.
2. Subjects aged 20 to 85 years.
3. Hemodialysis subjects with chronic renal failure and renal anemia in outpatient clinic currently on stable Eprex® treatment administered by intravenous injection (1 to 3 times per week) for at least 3 months prior to randomization.

Main Exclusion Criteria:

1. Maintenance epoetin dose > 300 IU/kg per week.
2. Treatment with long-acting epoetin analogues.
3. Detectable anti-erythropoietin antibodies with clinical symptoms at screening visit, or history of Pure Red Cell Aplasia (PRCA).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2016-03; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Mean change in hemoglobin (Hb) levels | Baseline and the evaluation period (evaluation period: Week21-Week24)
Mean change in weekly epoetin dosage. between baseline and the evaluation period | Baseline and the evaluation period (evaluation period: Week21-Week24)
Adverse events (AEs): incidence and severity of all drug-related AEs | up to 52 weeks
Immunogenicity: occurrence of anti-erythropoietin antibody | up to 52 weeks